CLINICAL TRIAL: NCT04522401
Title: Prevention of the Loss of Autonomy in the Old People: Factors Favoring or Limiting the Respect of Recommendations
Brief Title: Performance Evaluation Platform for Seniors.
Acronym: PEPS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A01075-50 (RIPH3); 2018-A01075-50 (Other: ANSM)
Record Dates: First submitted 2020-07-22; First posted 2020-08-21 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Aging
Keywords: old people; gerontological assessment; loss of autonomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People aged 65 and over: People aged 65 and over who have had a gerontological evaluation "Bien vieillir" at the St-Etienne University Hospital Day Hospital.
  Interventions: Diagnostic Test: consultation: "Bien vieillir"

INTERVENTIONS:
Diagnostic Test: consultation: "Bien vieillir" — Patients will benefit from a multidisciplinary assessment including a geriatric assessment standardized by a geriatrician, an evaluation by a dietician, an evaluation by an occupational therapist. They will then be exposed to a personalized plan of care in the form of a recommendation.Then, patients will be followed at home to evaluate the implementation of their personalized care plan at 3 months of their assessment day, then at 6 and 9 months.

SUMMARY:
Monocentric prospective non-randomized observational study with subgroup analysis on the assessment of the day hospital at the Aging Biennial Hospital of Saint-Etienne.

DETAILED DESCRIPTION:
Monocentric prospective non-randomized observational study with subgroup analysis on the assessment of the day hospital at the Aging Biennial Hospital of Saint-Etienne.

The main objective is to investigate the factors limiting or encouraging adherence to recommendations in a population aged over 65, fragile or pre-fragile, autonomous and living at home or in a shelter.

Patients will benefit from a multidisciplinary assessment including a geriatric assessment standardized by a geriatrician, an evaluation by a dietician, an evaluation by an occupational therapist. They will then be exposed to a personalized plan of care in the form of a recommendation.

Patients will be followed at home to evaluate the implementation of their personalized care plan at 3 months of their assessment day at the day hospital, then at 6 and 9 months. The study will take place over a period of approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Person affiliated or entitled to a social security scheme
* People aged 65 and over who participated in a consultation to age well at the day hospital of the St-Etienne university hospital during the study period.
* Elderly people who received an information about the study and who co-signed, with the investigator, a consent to participate in the study

Exclusion Criteria:

* Seniors who refused to participate
* Elderly people under legal protection measures
* Severe cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: seniors who have had a gerontological assessment
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
rate of implementation of recommendations concerning mobility (adapted physical activity). | Months: 9
  This rate is the ratio between the number of mobility recommendations made at 9 months and the number initially recommended.
  Analysis by tracking sheet patient results.

SECONDARY OUTCOMES:
Overall rate of implementation of the recommendations at 9 months | Months: 9
  Analysis by tracking sheet patient results.
Satisfaction rate of the platform's users | Months: 9
  Analysis by qualitative interviews results.

CONTACTS AND LOCATIONS:
Overall Officials: Romain JUGAND, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No